CLINICAL TRIAL: NCT04454710
Title: The Efficacy of Pulsed Radiofrequency on the Saphenous Nerve in Osteoarthritic Chronic Knee Pain
Brief Title: Pulsed Radiofrequency and Osteoarthritic Chronic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Mohammad Alwardat, Postdoctoral fellowship, University of Rome Tor Vergata
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 144/18
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Pulsed Radiofrequency; Osteoarthritis, Knee; Knee Pain Chronic; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Pulsed Radiofrequency (Active Comparator): The participant will receive real pulsed radiofrequency for 2 minutes at a frequency of 2 pulses per second (2Hz) while lie in the supine position with their leg of interest partially flexed about 45 degrees and externally rotated. The full procedure will take eight minutes, composed of four sessions of 2 minutes in which the temperature was maintained below 42°C.
  Interventions: Device: Pulsed Radiofrequency
- Sham Pulsed Radiofrequency (Sham Comparator): Identical to the real pulsed radiofrequency, except the participants will only receive the initial 2 seconds of ramp-up, after which the device will switch-off for the rest of the session and will turn-on again at the end of the session.
  Interventions: Device: Pulsed Radiofrequency

INTERVENTIONS:
Device: Pulsed Radiofrequency — Pulsed radiofrequency is a novel therapeutic modality with many potential applications in pain management.

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of pulsed radiofrequency of the saphenous nerve in the treatment of pain due to knee osteoarthritis (OA). The investigators will conduct real pulsed radiofrequency or sham, over the saphenous nerve during 4 separate sessions. The investigators will evaluate pain intensity, quality of life, function, and disability via clinical validated scales.

The research question is whether pulsed radiofrequency can lessen knee pain and improve function and quality of life in patients with chronic knee pain due OA.

It is hypothesized, that less knee pain and improved function, and quality of life after the pulsed radiofrequency sessions.

DETAILED DESCRIPTION:
Osteoarthritis (OA) affects 10% of the population over 60 years of age each year, with an increasing incidence related to population aging. This disease costs 1-2.5% of GDP on average in Europe when combining direct and indirect costs: it is therefore the 9th leading cause of disability adjusted life years. The knee is the most commonly affected joint, for which there is no treatment able to stop joint degeneration as of today: common treatment regimens include pharmacological therapy, joint infiltrations, neuromodulation techniques, and total knee arthroplasty when indicated. However, each patient responds differently and therefore necessitates a tailored approach.

Pulsed radiofrequency (PRF), a neuromodulating technique that potentiates the descending analgesic pathway by avoiding Wallerian degeneration, has as of today been targeted intraarticularly or to the genicular nerves, yielding unreliable results in both cases, perhaps due to small samples, lack of long term follow ups, and absence of control groups.

The goal of this study is to explore the efficacy and safety of PRF on the saphenous nerve, an exclusively sensory nerve that is responsible for pain perception on the medial surface of the lower limb, often associable with OA. In particularly, the investigators will evaluate the effect of PRF on pain reduction, function, disability, and quality of life in patients with knee OA.

This study will include 20 participants suffering from knee OA, and the participants will enroll if infiltrating their saphenous nerve with 2mL of 2% lidocaine reduces their Numeric Pain Rating Scale (NRS) pain perception by at least 60%.

The participants will be allocated consecutively to randomization as an intervention order using the tool from the randomization.com website (Dallal GE, http://www.randomization.com). The investigators will use the second generation suggested for crossover studies. The participants will be randomized into a PRF sham control group or a real PRF group and the investigators will follow up at 2 weeks (T1), 1 month (T2), 3 months (T3), and 6 months (T4) by acquiring their NRS, Oxford Knee Score, and SF-36 questionnaire. After 6 months, the participants will be crossed-over and the follow-up method will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Chronic knee pain (present for at least 6 months), of moderate-severe intensity (assessed by NRS => 6), not responsive to conservative treatments (physiotherapy, oral analgesics).
* Diagnosis of knee osteoarthritis confirmed by instrumental investigation (X-ray and/or MRI) and Oxford Knee Score = <35.
* Positivity to the diagnostic block of no. saphenous (defined as a reduction of at least 50% of the NRS score).
* If the patient is taking opioids or other morphine equivalents, the dosage should not be changed within 3 months prior to the study enrollment visit.

Exclusion Criteria:

* Body Mass index > 40 kg /m2
* History of systemic inflammatory disease, uncontrolled diabetes mellitus, neoplastic pathology, coagulopathy
* Previous knee replacement implant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in Pain severity | Measured at baseline and immediately after the intervention]
  Changes in Pain severity will be measured by Numeric Pain Rating Scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable").

SECONDARY OUTCOMES:
Changes in Health related quality-of -life | Measured at baseline and immediately after the intervention]
  Changes in quality of life will be measured by SF-36. The Italian version of SF-36 will used to understand the health related quality-of -life of the participants over the past four weeks. The eight health concepts: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions will be searched. These outcomes will be grouped as physical component summary and mental component summary. The norm data is 0-100, the health related quality of life is increases as the scores are increased. The average score is 50.
Changes in in knee function and pain | Measured at baseline and immediately after the intervention]
  Changes in in knee function and pain will be measured by Oxford Knee Score. The Oxford Knee Score questionnaire consists of 12 questions that cover function and pain of the knee. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome Tor Vergata, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang W, Doherty M, Peat G, Bierma-Zeinstra MA, Arden NK, Bresnihan B, Herrero-Beaumont G, Kirschner S, Leeb BF, Lohmander LS, Mazieres B, Pavelka K, Punzi L, So AK, Tuncer T, Watt I, Bijlsma JW. EULAR evidence-based recommendations for the diagnosis of knee osteoarthritis. Ann Rheum Dis. 2010 Mar;69(3):483-9. doi: 10.1136/ard.2009.113100. Epub 2009 Sep 17. PMID 19762361
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, part I: critical appraisal of existing treatment guidelines and systematic review of current research evidence. Osteoarthritis Cartilage. 2007 Sep;15(9):981-1000. doi: 10.1016/j.joca.2007.06.014. Epub 2007 Aug 27. PMID 17719803
- [Background] Kapoor R, Adhikary SD, Siefring C, McQuillan PM. The saphenous nerve and its relationship to the nerve to the vastus medialis in and around the adductor canal: an anatomical study. Acta Anaesthesiol Scand. 2012 Mar;56(3):365-7. doi: 10.1111/j.1399-6576.2011.02645.x. PMID 22335278
- [Background] Carlino E, Piedimonte A, Benedetti F. Nature of the placebo and nocebo effect in relation to functional neurologic disorders. Handb Clin Neurol. 2016;139:597-606. doi: 10.1016/B978-0-12-801772-2.00048-5. PMID 27719874
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Castelnuovo G, Giusti EM, Manzoni GM, Saviola D, Gabrielli S, Lacerenza M, Pietrabissa G, Cattivelli R, Spatola CAM, Rossi A, Varallo G, Novelli M, Villa V, Luzzati F, Cottini A, Lai C, Volpato E, Cavalera C, Pagnini F, Tesio V, Castelli L, Tavola M, Torta R, Arreghini M, Zanini L, Brunani A, Seitanidis I, Ventura G, Capodaglio P, D'Aniello GE, Scarpina F, Brioschi A, Bigoni M, Priano L, Mauro A, Riva G, Di Lernia D, Repetto C, Regalia C, Molinari E, Notaro P, Paolucci S, Sandrini G, Simpson S, Wiederhold BK, Gaudio S, Jackson JB, Tamburin S, Benedetti F. What Is the Role of the Placebo Effect for Pain Relief in Neurorehabilitation? Clinical Implications From the Italian Consensus Conference on Pain in Neurorehabilitation. Front Neurol. 2018 May 18;9:310. doi: 10.3389/fneur.2018.00310. eCollection 2018. PMID 29867723
- [Background] Gupta A, Huettner DP, Dukewich M. Comparative Effectiveness Review of Cooled Versus Pulsed Radiofrequency Ablation for the Treatment of Knee Osteoarthritis: A Systematic Review. Pain Physician. 2017 Mar;20(3):155-171. PMID 28339430
- [Background] Herman DC, Vincent KR. Saphenous Nerve Block for the Assessment of Knee Pain Refractory to Conservative Treatment. Curr Sports Med Rep. 2018 May;17(5):146-147. doi: 10.1249/JSR.0000000000000480. No abstract available. PMID 29738318
- [Background] Kesikburun S, Yasar E, Uran A, Adiguzel E, Yilmaz B. Ultrasound-Guided Genicular Nerve Pulsed Radiofrequency Treatment For Painful Knee Osteoarthritis: A Preliminary Report. Pain Physician. 2016 Jul;19(5):E751-9. PMID 27389118
- [Derived] Carpenedo R, Al-Wardat M, Vizzolo L, Germani G, Chine E, Ridolfo S, Dauri M, Natoli S. Ultrasound-guided pulsed radiofrequency of the saphenous nerve for knee osteoarthritis pain: a pilot randomized trial. Pain Manag. 2022 Mar;12(2):181-193. doi: 10.2217/pmt-2021-0035. Epub 2021 Aug 25. PMID 34431329